CLINICAL TRIAL: NCT06894342
Title: Ultrasonographic Evaluation of the Effect of Occlusal Splint Treatment on Masseter Muscle Thickness in Children With Sleep Bruxism:A Clinical Pilot Study
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, zeynepbetul, Assoc. Prof. Dr., Ankara Yildirim Beyazıt University
Other Study IDs: AYBU-DHF-ZBA-01
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Bruxism, Sleep
Keywords: bruxism; child; USG; masseter muscle; occlusal splint
MeSH Terms: conditions — Sleep Bruxism; Bruxism | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Patients between the ages of 7 and 12, with mixed dentition, class I occlusion and diagnosed with probable bruxism
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Ultrasonographic evaluation of the masseter muscle

SUMMARY:
The aim of this study was to evaluate the effectiveness of occlusal splint in pediatric bruxist patients by ultrasonic measurements of masseter muscle thickness and pain perception.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effectiveness of occlusal splint by ultrasonographic measurements of masseter muscle thickness and pain perception in a group of pediatric bruxist patients. The study included patients aged 7 to 12 years, all in the mixed dentition period, with class I occlusion and diagnosed with probable bruxism. A 2 mm thick soft occlusal splint was prepared for each patient. Ultrasonic measurements were used to assess the thickness of the masseter muscle (MMT) at baseline, one, two and three months.Visual Analog Scale (VAS) was also used to record subjective pain measurements. Repeated-measures ANOVA and Friedman test were used in the statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of tooth clenching or grinding when sleeping at night or during the day, including headaches in the morning, as reported by parents during anamnesis.
* Attrition-type tooth wear, as well as discomfort, fatigue, and/or pain in the jaw muscles when palpated during a clinical examination. The clinical diagnosis of attrition was based on the following findings:

  * Shiny and flat facets.
  * The enamel and dentin wear at the same pace.
  * Wear patterns on opposing teeth's occlusal surfaces.
  * Possible breakage of cusps or restorations.
  * Impressions on the cheeks, tongue, or lips.

Exclusion Criteria:

* Children with any chronic/systemic/psychological disease, presence of TMD symptoms, lack of posterior teeth that may cause unilateral chewing, use of any medication that may affect muscle activity, dental malocclusions (any skeletal jaw problems in anteroposterior and vertical dimensions) and ongoing orthodontic treatment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients between the ages of 7 and 12, with mixed dentition, class I occlusion and diagnosed with probable bruxism
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
muscle thickness measurement | from the beginning to the third month
  Masseter muscle thicknes was measured from a single position at the thickest part of the muscle, close to the occlusal plane and midway between the zygomatic arch and the gonial angle. Masseter muscle thicknes was evaluated bilaterally, in both the relaxed and contracted (maximum biting) positions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No